CLINICAL TRIAL: NCT06617455
Title: Phase 2 Randomized, Cross-over Trial of Fezolinetant for Treatment of Vasomotor Symptoms in Patients Taking Endocrine Therapy (VEnT)
Brief Title: Fezolinetant for the Improvement of Vasomotor Symptoms in Breast Cancer Patients Taking Endocrine Therapy, VENT Trial
Acronym: VEnT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: The Breast Cancer Research Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: UMCC 2024.059; NCI-2024-06543 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HUM00256706 (Other: University of Michigan)
Record Dates: First submitted 2024-09-24; First posted 2024-09-27 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Breast Ductal Carcinoma In Situ; Localized Breast Carcinoma
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating | interventions — Specimen Handling; fezolinetant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All study drug will be blinded to the patients, the study investigators, and the study coordinators to ensure masking of the treatments. The statistician and the study investigators will remain blinded until the study database is locked. The only study personnel that will not be blinded are the research pharmacy staff in order to facilitate randomization codes and treatment delivery, and in case emergency unblinding is required.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (fezolinetant, placebo) (Experimental): Patients receive fezolinetant PO QD for 28 days in the absence of unacceptable toxicity. Patients then go through a washout period and take no study medication for the next 14 days. Following the washout, patients receive placebo PO QD for 28 days in the absence of unacceptable toxicity. Patients undergo collection of blood samples throughout the study.
  Interventions: Procedure: Biospecimen Collection; Drug: Fezolinetant; Drug: Placebo Administration; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (placebo, fezolinetant) (Experimental): Patients receive placebo PO QD for 28 days in the absence of unacceptable toxicity. Patients then go through a washout period and take no study medication for the next 14 days. Following the washout, patients receive fezolinetant PO QD for 28 days in the absence of unacceptable toxicity. Patients undergo collection of blood samples throughout the study.
  Interventions: Procedure: Biospecimen Collection; Drug: Fezolinetant; Drug: Placebo Administration; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Fezolinetant — Given PO
Drug: Placebo Administration — Given PO
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial tests how well fezolinetant works in improving vasomotor symptoms (VMS) in breast cancer patients taking endocrine therapy (ET). Anti-hormone treatments are effective for lowering the risk of breast cancer but can cause bothersome VMS, such as hot flashes and night sweats. Fezolinetant inhibits the activity of the neurokinin type 3 receptor and has shown activity against VMS in postmenopausal women. Taking fezolinetant may work well at improving VMS in breast cancer patients taking ET.

ELIGIBILITY:
Inclusion Criteria:

* Female subject aged ≥ 18 years
* Taking endocrine therapy (tamoxifen, anastrozole, exemestane, or letrozole) for adjuvant treatment of stage 1-3 breast cancer or for chemoprevention (breast ductal carcinoma in situ [DCIS] or high risk)
* Planning to take the same endocrine therapy for at least 10 weeks after study drug initiation
* Report 28 or more VMS episodes, at least some of which are severe or bothersome, during the 7-day screening period
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2 x upper limit of normal (ULN) within 28 days prior to randomization
* Total bilirubin < 2 x ULN within 28 days prior to randomization
* Completion of chemotherapy, if given. Concurrent use of gonadotropin releasing hormone agonist (GnRHa) therapy, anti-HER2 therapy, bisphosphonate therapy, poly adenosine diphosphate-ribose polymerase (PARP) inhibitor therapy, and abemaciclib therapy is permitted
* Patients receiving treatment with selective serotonin reuptake inhibitor (SSRIs), serotonin and norepinephrine reuptake inhibitor (SNRIs), gabapentinoids, clonidine, or oxybutynin must have been taking a stable dose for at least 30 days prior to enrollment if they plan to continue the drug during study participation, and willing to remain on the treatment for the duration of study participation. If they do not plan to take the medication during study participation, they should stop the medication at least 7 days before the start of the VMS screening period
* Patients taking over-the-counter supplements or herbal medications for treatment of VMS must stop the medication at least 7 days before the start of the VMS screening period
* Able to self-complete questionnaires in English
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines
* For women of childbearing potential, participants must agree to use an effective contraceptive method during protocol therapy and for 3 months following completion of protocol therapy with details provided as a part of the consent process and must have a negative pregnancy test at screening. In addition to routine contraceptive methods, "effective contraception" also includes refraining from sexual activity that might result in pregnancy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) including hysterectomy, bilateral oophorectomy, and bilateral tubal ligation/occlusion

Exclusion Criteria:

* Metastatic breast cancer
* Prior treatment with fezolinetant
* Known severe renal disease (estimated glomerular filtration rate [eGFR] less than 30 mL/min/1.73 m^2)
* Known cirrhosis
* Pregnant or breast feeding, or plan to become pregnant during the study period or within 3 months of completing study medication
* Concomitant use of CYP1A2 inhibitors, including but not limited to fluvoxamine, ciprofloxacin, cimetidine, citalopram, and ribociclib
* Concomitant use of systemic or transdermal estrogen products
* Known allergy or hypersensitivity to fezolinetant or any of the excipients in the medication
* Unable to take oral medications
* Any medical condition that would interfere with the absorption of study medication. Prior gastric bypass is permitted
* Concurrent medical disease that could confound or interfere with evaluation of VMS
* Patients with a prior or concurrent malignancy whose natural history or treatment, in the opinion of the treating investigator, has the potential to interfere with the safety or efficacy assessment of the investigational regimen
* Patients who are participating concurrently in another interventional study (actually receiving a study medication) or participated in an interventional study within 30 days prior to screening or received any investigational drug within 30 days or within 5 half-lives prior to screening, whichever is longer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in frequency of vasomotor symptoms (VMS) | Baseline to day 71
  Will perform an intent-to-treat analysis. The mean change in frequency of VMS with 4 weeks of fezolinetant versus placebo will be reported with the corresponding 95% confidence interval. Initial analysis will use a paired t-test of the mean change in frequency of VMS with 4 weeks of treatment with drug and placebo. Follow up analyses will use a linear mixed effects model (with any transformation needed for assumptions to be met) with random intercept that considers the repeated measurements, possible sequence, period, and carryover effects.

SECONDARY OUTCOMES:
Change of the severity of VMS | Baseline to day 71
  The mean change of the severity of VMS, as assessed with the hot flash log, with 4 weeks of fezolinetant versus placebo. Will perform an intent-to-treat analysis. Will be reported with corresponding 95% confidence intervals. Initial analysis will use a paired t-test of the mean change in severity of VMS from baseline to week 4 between drug and placebo. Follow up analyses will use a linear mixed effects model (with any transformation needed for assumptions to be met) with random intercept that considers the repeated measurements, possible sequence, period, and carryover effects.
Change of the hot flash score | Baseline to day 71
  The mean change of the hot flash score, as assessed with the hot flash log and calculated by multiplying VMS frequency by severity, with 4 weeks of fezolinetant versus placebo. Will perform an intent-to-treat analysis. Will be reported with corresponding 95% confidence intervals. Initial analysis will use a paired t-test of the mean change in hot flash score from baseline to week 4 between drug and placebo. Follow up analyses will use a linear mixed effects model (with any transformation needed for assumptions to be met) with random intercept that considers the repeated measurements, possible sequence, period, and carryover effects.
Change of the Menopause-Specific Quality of Life (MENQOL) hot flash subscore | Baseline to day 71
  The mean change of the MENQOL hot flash subscore with 4 weeks of fezolinetant versus placebo. Will perform an intent-to-treat analysis. Will be reported with corresponding 95% confidence intervals. Initial analysis will use a paired t-test of the mean change in MENQOL hot flash subscore from baseline to week 4 between drug and placebo. Follow up analyses will use a linear mixed effects model (with any transformation needed for assumptions to be met) with random intercept that considers the repeated measurements, possible sequence, period, and carryover effects.
Patient Global Impression of Change (PGIC) for hot flashes and night sweats | Baseline to day 71
  The mean PGIC for hot flashes and for night sweats after 4 weeks of fezolinetant versus placebo. Will perform an intent-to-treat analysis. Will be reported with corresponding 95% confidence intervals. Initial analysis will use a paired t-test of PGIC score from baseline to week 4 between drug and placebo. Follow up analyses will use a linear mixed effects model (with any transformation needed for assumptions to be met) with random intercept that considers the repeated measurements, possible sequence, period, and carryover effects.
Change of the Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance | Baseline to day 71
  The mean change of the PROMIS Sleep Disturbance T score with 4 weeks of fezolinetant versus placebo. Will perform an intent-to-treat analysis. Will be reported with corresponding 95% confidence intervals. Initial analysis will use a paired t-test of the mean change in PROMIS Sleep Disturbance from baseline to week 4 between drug and placebo. Follow up analyses will use a linear mixed effects model (with any transformation needed for assumptions to be met) with random intercept that considers the repeated measurements, possible sequence, period, and carryover effects.
Incidence of adverse events | Baseline through 30 days after the last dose of study treatment
  Safety will be assessed throughout the trial and adverse events during the 10 weeks of study participation will be reported using descriptive statistics for fezolinetant and for placebo. Assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Norah L Henry, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Rogel Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
participant demographics and patient-reported outcomes data will be available to researchers upon reasonable request
Supporting Information: Study Protocol, SAP
Time Frame: researchers can request data once the primary analysis has been published
Access Criteria: deidentified data will be available to researchers upon reasonable request

REFERENCES:
- See also: Related Info — https://UMHealthResearch.org/studies/HUM00256706